CLINICAL TRIAL: NCT00906165
Title: The Role of Immediate Provisional Restorations on Bone Level Implants. A Randomised, Single Blind Controlled Clinical Trial
Brief Title: The Role of Immediate Provisional Restorations on Bone Level Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR 05/07
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Jaw, Edentulous, Partially
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1- Immediately provisionalized (Active Comparator): The Straumann® Bone Level SLActive Implant (4.1mm diameter) will be immediately provisionalized upon placement, i.e. impressions will be taken directly after implant installation in order to fabricate screw-retained resin crowns within 48 hours after implant placement. At 16 weeks, the final prosthetic reconstruction will be performed according to the standard procedure for single crown restoration.
  Interventions: Device: Straumann® Bone Level SLActive Implant (4.1mm diameter)
- 2- Delayed Loading (Active Comparator): The Straumann® Bone Level SLActive Implant (4.1mm diameter) will not be immediately provisionalized, instead there will be delayed implant loading. i.e. the patient will receive a removable prosthesis if necessary and the impressions for the final restoration will be taken 12-14 weeks after implant installation. At 16 weeks, the final prosthetic reconstruction will be performed according to the standard procedure for single crown restoration.
  Interventions: Device: Straumann® Bone Level SLActive Implant (4.1mm diameter)

INTERVENTIONS:
Device: Straumann® Bone Level SLActive Implant (4.1mm diameter) — Straumann® Bone Level Implants will be placed in healed alveolar ridge (at least 8 weeks post extraction). Implants in Arm 1 will be immediately provisionalized. Implants in Arm 2 will not be immediately provisionalized. Implants in both Arms will be loaded at 16 weeks (final prosthetic reconstruction will be performed according to the standard procedure for single crown restoration)

SUMMARY:
The study is designed to evaluate the clinical and radiographic outcomes of Straumann® Bone Level Implant SLActive placed in healed alveolar ridge (at least 8 weeks post extraction) and immediately provisionalised versus the same type of implants placed in healed alveolar ridge but not provisionalised. In both cases the implants will be loaded at 16 weeks (final restorations). The outcomes will be evaluated over a 2-year period.

DETAILED DESCRIPTION:
This is a prospective, randomised, controlled, single blind, and single center study. The total study duration for each patient should be 24 months.

Straumann Bone Level Ø 4.1 mm SLActive implants will be placed for single tooth replacement, followed by either immediate provisional prosthetic loading or no provisionalised. The final prosthetic loading is made at 16 weeks after implant loading. The implant length will be selected according to the clinical indication of the site based on previous radiographic evaluation.

In total 11 visits per patient are scheduled in this study. Bone level changes, implant success and survival rate, soft tissue changes, aesthetic outcome and adverse events (AEs) will be assessed.

The study devices are CE- (Conformité Européenne, meaning European Conformity) marked products.

One center in the United Kingdom will participate.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria

  * Males and females, age 18 to 75 years of age (the subjects should be legally able to give informed consent to the procedure; age limitation is also present to avoid inclusion of subjects with incomplete cranio-facial growth).
  * Absence of relevant medical conditions. Patients with contributing medical history in which any elective oral surgical intervention would be contraindicated should be excluded. In particular patients with uncontrolled or poorly controlled diabetes, or unstable or life threatening conditions should be excluded.
  * Absence of uncontrolled or untreated periodontal disease.
  * Absence of untreated caries lesions.
  * Patient in good medical and psychological health as documented by self assessment
  * Patient's availability for follow-up according to the protocol.
* Local inclusion criteria

  * A single tooth replacement is required in the incisor, canine, pre-molar and first molar region. Multiple-implant restorations (non adjacent to the test implant) can be performed during the study (not to be included as test implants).
  * at least 8 weeks post extraction where the soft tissues of the socket have healed
  * Presence of at least one adjacent tooth
  * Presence of adequate native bone to achieve primary stability

Exclusion Criteria:

* General exclusion criteria

  * Patients who have any known diseases (not including controlled diabetes mellitus), infections or recent surgical procedures within 30 days of study initiation.
  * Female patients who are pregnant or lactating or of child bearing potential not using acceptable methods of birth control (hormonal, barriers or abstinence).
  * Patients who are on chronic treatment (i.e., two weeks or more) with any medication known to affect oral status (e.g., phenytoin, dihydropyridine, calcium antagonists, cyclosporine) within one month of baseline visit.
  * Patients who are on concomitant anticoagulant therapy of warfarin (coumadine), clopidogrel, ticlopidine or once daily aspirin of more than 81 mg.
  * Patients who knowingly have HIV or Hepatitis.
  * Physical handicaps that would interfere with the ability to perform adequate oral hygiene.
  * Patients who have undergone administration of any investigational drug within 30 days of study initiation.
  * Alcoholism or chronically drug abuse causing systemic compromisation.
  * Patients who are heavy smokers (>10/cigarettes per day).
  * Patients suffering from a known psychological disorder.
  * Patients who have limited mental capacity or language skills such that study information cannot be understood, informed consent cannot be obtained or simple instructions cannot be followed.
  * Exclude patients with BOP > 30% at the completion of the pre-treatment phase.
* Local exclusion criteria

  * Exclude experimental sites with inadequate bone availability where initial stability of the implant cannot be achieved or extended augmentation procedures and/ or sinus nasal lift are required.
  * History of local radiation therapy.
  * Presence of severe oral lesions.
  * Severe bruxism or clenching habits
  * Patients with lack of posterior occlusion and severely reduced vertical dimension of occlusion
  * Patients presenting clinical and radiological signs and symptoms of maxillary sinus disease in the implant area.
  * Patients presenting an acute endodontic lesion in the neighboring areas to the experimental procedure (sites with presence of an asymptomatic chronic lesion are eligible)
  * Plaque score > 30%

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-06; Primary Completion 2011-11 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Donos, Prof. Dr., Principal Investigator — Eastman Dental Institute
Locations (1):
- Eastman Dental Institute, University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1- Immediately Provisionalized | 2- Delayed Loading
Started | 14 | 14
Completed | 10 | 14
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1- Immediately Provisionalized | 2- Delayed Loading | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 1 | 0 | 1
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 42.1 [39.1 to 49.5] | 47.9 [41.5 to 52.2] | 45.3 [39.4 to 52.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Bone Level Change at the Mesial and Distal of the Implants Between Baseline and One Year Post Treatment
Description: The primary parameter derives from the subtraction of mesial and distal bone level linear x-ray measurements at baseline and one year after implant placement. The distance between the alveolar bone at the level of the first radiographic bone contact with the implant surface and the shoulder of the implant will be measured to the closest 0.1mm at the mesial and distal surfaces of all implants, on digitized standardized peri-apical x-rays using an image analysis computer program.
Time Frame: between baseline and one year post treatment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 1- Immediately Provisionalized | 2- Delayed Loading
Number analyzed (Participants) | 10 | 14
mm | 0.73 (0.83) | 0.22 (0.46)

2. Secondary Outcome: Number of Participants With Survival Rate of the Implants at 12 and 24 Months
Description: The survival rate of the implants is presented as a cumulative survival rate at 1 year and 2 years post-implant placement.
Time Frame: 1 year and 2 years after implant placement
Population: Survival rate of the implants at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 1- Immediately Provisionalized | 2- Delayed Loading
Number analyzed (Participants) | 14 | 14
Participants
  No. of participants w. implant survival of 12mts | 14 | 14
  No. of participants w. implant survival of 24mts | 14 | 14

3. Secondary Outcome: No. of Participants With Complications of the Implant and Implant Overstructure at 24 Months
Description: No of participants with prosthetic related complications and with implant failures are described after 24 months
Time Frame: 2 years after implant placement
Measure: Number; unit: participants
Arm/Group | 1- Immediately Provisionalized | 2- Delayed Loading
Number analyzed (Participants) | 14 | 14
participants
  Number of prosthetic related complications | 1 | 1
  Number of implant failures | 0 | 0

4. Secondary Outcome: Probing Pocket Depth
Description: The Probing Pocket Depth around the implants will be measured using a UNC-15 probe with light probing force (0.2N) at the post-implant time-points specified. Differences between the Outcome Measure time points will be displayed. Baseline is 16 weeks (loading of implants)
Time Frame: Recorded at 16 weeks, 6, 12, and 24 months after implant placement
Population: Difference of Probing Pocket Depth (PPD) between 16 weeks (loading) and 6 months, 12 months and 24 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 1- Immediately Provisionalized | 2- Delayed Loading
Number analyzed (Participants) | 10 | 14
mm
  PPD difference 16weeks-6months | -0.3 (0.5) | -0.5 (0.7)
  PPD difference 16weeks-12 months | -0.4 (0.8) | -0.7 (0.9)
  PPD difference 16weeks-24 months: number analyzed (Participants) | 10 | 13
  PPD difference 16weeks-24 months | -0.1 (0.7) | -0.8 (1.0)

5. Secondary Outcome: Gingival Recessions (REC)
Description: The gingival recessions around the implants are recorded at the above-specified timepoints after implant placement, using a UNC-15 probe. Differences between the Outcome Measure time points will be displayed. Baseline is 16 weeks (loading of implants)
Time Frame: Recorded at 16 weeks, 6, 12 and 24 months after implant placement
Population: Patient 218 discontinued the study after 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 1- Immediately Provisionalized | 2- Delayed Loading
Number analyzed (Participants) | 10 | 14
mm
  REC difference 16weeks-6months | 0.1 (0.2) | 0.4 (0.3)
  REC difference 16weeks-12months | 0.2 (0.3) | 0.5 (0.4)
  Recession at 24 months: number analyzed (Participants) | 10 | 13
  Recession at 24 months | 0.2 (0.4) | 0.5 (0.3)

6. Secondary Outcome: Number of Participants With Soft Tissue Changes Assessed by Papilla Fill Index
Description: Soft tissue changes: mesial and distal gingival papilla dimensions assessed by Papilla Fill Index (PFI, Jemt 1997) and the Pink Aesthetic Score (PES, Furhauser 2005) will be recorded at the post-implant placement timepoints specified above.
Time Frame: Recorded at 12 and 24 months after implant placement
Population: Patient 218 discontinued the study after 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 1- Immediately Provisionalized | 2- Delayed Loading
Number analyzed (Participants) | 10 | 14
Participants
  PFI 12m: 0=absent papilla | 0 | 0
  PFI 12m: 1=incomplete Papilla 1/3 of full | 2 | 2
  PFI 12m: 2=incomplete papilla 2/3 of full | 6 | 6
  PFI 12m: 3=complete papilla | 2 | 6
  PFI 24m: 0=absent papilla: number analyzed (Participants) | 10 | 13
  PFI 24m: 0=absent papilla | 0 | 0
  PFI 24m: 1=incomplete Papilla 1/3 of full | 1 | 0
  PFI 24m: 2=incomplete papille 2/3 of full | 5 | 7
  PFI 24m: 3=complete papilla | 4 | 6

7. Secondary Outcome: Adverse Events
Description: Adverse Events (AE) and Serious Adverse Events (SAE) will be assessed and followed up throughout the study duration
Time Frame: From randomization to 2 years after implant placement
Population: Patient 218 discontinued the study after 12 months
Measure: Number; unit: events
Arm/Group | 1- Immediately Provisionalized | 2- Delayed Loading
Number analyzed (Participants) | 14 | 14
events
  AE at 12 months | 15 | 22
  AE 12 - 24 months: number analyzed (Participants) | 14 | 13
  AE 12 - 24 months | 7 | 6

8. Secondary Outcome: Soft Tissue Changes, Pink Aesthetic Score
Description: Soft tissue changes: the Pink Aesthetic Score (PES, Furhauser 2005) will be recorded at the post-implant placement timepoints specified above.
  The PES index includes assessment of seven variables and each variable is measured with a 2, 1, or 0 score with 2 being the best and 0 being the poorest score. Based on its definition the PES is a cumulative score with 14 being the best and 0 the worst.
Time Frame: Recorded at 12 and 24 months after implant placement
Population: Patient 218 discontinued the study after 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1- Immediately Provisionalized | 2- Delayed Loading
Number analyzed (Participants) | 14 | 14
score on a scale
  PES at 12 months: number analyzed (Participants) | 9 | 14
  PES at 12 months | 11.4 (1.2) | 11.6 (1.0)
  PES at 24 months: number analyzed (Participants) | 9 | 13
  PES at 24 months | 11.6 (1.3) | 11.6 (0.7)

ADVERSE EVENTS:
Arm/Group | 1- Immediately Provisionalized | 2- Delayed Loading
Serious Adverse Events (participants affected / at risk) | 0/14 | 2/14
Other Adverse Events (participants affected / at risk) | 9/14 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1- Immediately Provisionalized (N=14) | 2- Delayed Loading (N=14)
Atrial flutter (Cardiac disorders) | 0 | 1 — Hospitalization
Cardiac ablation (Cardiac disorders) | 0 | 1 — Hospitalization
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1- Immediately Provisionalized (N=14) | 2- Delayed Loading (N=14)
Implant or procedure related complications (Product Issues) | 3 | 1
Prosthetic related complication (Product Issues) | 2 | 7 — any Event related to the prosthetic procedures
clinical conditions (General disorders) | 4 | 4 — Condition found during visit. Events not related to device or procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days